CLINICAL TRIAL: NCT06536881
Title: Gut Microbiome, Adverse Effects, and Markers Through MEtabolic Reprogramming (GAMMER) Study in Early Stage Breast Cancer Receiving Chemotherapy
Brief Title: Gut Microbiome, Adverse Effects, and Markers Through MEtabolic Reprogramming
Acronym: GAMMER
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: The Commonwealth Fund (Other); Maryland Cigarette Restitution Fund (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: J2362; IRB00390964 (Other: JHM IRB)
Record Dates: First submitted 2024-07-31; First posted 2024-08-05 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Breast Cancer; Early-stage Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Angptl4 protein, mouse

STUDY DESIGN:
Intervention Model Description: Participants undergo a trial of 24-hour water only fasting before starting chemotherapy. At least one successful 24-hour fast is required. A total of 3 trials can be attempted. Participants can also progressively increase by 12 hours each week as tolerated or to a max of 48 hours. If a participant is unable to maintain at least a 24-hour fast during the study, participation in this study will end. Once the tolerated fasting time is established, this will be the starting fasting regimen used for Cycle 1 of 4 of the scheduled chemotherapy.
  Investigators also aim to understand the impact of fasting on quality of life, inflammatory markers, and the bacteria in the gut. Participants will complete surveys weekly, blood samples for research and fasting labs with each cycle of chemotherapy (at 4 different time points). Investigators will also collect research bloods at baseline, stool samples 3 times in the study: baseline, and after fasting interventions for Cycle 1 and 3.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fasting prior to chemotherapy (Experimental): Prior to chemotherapy administration, a trial of a 24-hour water-only fast will be conducted; at least 1 successful 24-hour fast is required to proceed with the fasting intervention during chemotherapy. A total of 3 trials is allowed (for a maximum of 48 hours fasting).
  Interventions: Behavioral: Fasting

INTERVENTIONS:
Behavioral: Fasting — The dietician will review the patient's chemotherapy schedule, and confirm the fasting window (as windows may be 24, 26 or 48 hours; and chemotherapy start times can vary from patient to patient).

SUMMARY:
This research is being done to test the feasibility of 24-48 hours of water-only fasting to improve delivery of 4 cycles of chemotherapy in those receiving breast cancer treatment either before or after surgery.

DETAILED DESCRIPTION:
Breast cancer is the most common cancer diagnosed among women worldwide. Many women diagnosed with early stage breast cancer (ESBC) will receive systemic therapy consisting of cytotoxic chemotherapy. As therapy-related toxicities are the most common reason for non-completion or dose reduction of chemotherapy, new strategies are needed to mitigate adverse effects. Preclinical studies show that fasting can prevent toxic effects of oxidative stress and chemotherapy without causing chronic weight loss via modulation of key oncogenic pathways. A few studies in women with breast cancer have demonstrated that fasting around chemotherapy is safe and has the same or fewer expected toxicities, although the underlying biological mechanisms for these findings is unknown. A better understanding of the mechanistic underpinnings of fasting interventions can lead to future interventions to enhance tolerability of chemotherapy and ultimately, maintaining intended chemotherapy dosing and schedule.

The primary objective of this study is to determine the feasibility of water-only fasting during chemotherapy (standard of care Taxotere and Cyclophosphamide (TC) every 3 weeks for 4 cycles or dose dense doxorubicin and cyclophosphamide (ddAC) every 2 weeks for 4 cycles) in 30 patients with early stage breast cancer. Concomitant human epidermal growth factor 2 (HER2) therapy is allowed. The investigators designed a bed-to-bench feasibility study called the Gut microbiome, Adverse effects, and Markers through MEtabolic Reprogramming (GAMMER) study. Feasibility will be evaluated by the proportion of participants with self-reported adherence to the fasting regimen. The investigators will consider the fasting intervention to be feasible if there is evidence that at least 70% of patients (corresponding with 24 out of 30 patients) adhere to the intervention for at least 3 of 4 cycles of chemotherapy.

Prior to chemotherapy, patients will undergo a dose finding for fasting. A minimum of one successful 24 hour fast is required during this. A maximum of three trials is allowed. Participants have the option to progressively increase the fasting window by 12 hours each week as tolerated or to a maximum of 48 hours). Patients who are unable to adhere to at least a 24 hour fast during the dose finding phase will be replaced. Once patients have a fasting dose established, this will be the starting dose used for Cycle 1 of 4 of scheduled chemotherapy.

The investigators also aim to understand the impact of short-term fasting on quality of life, as well as key cytokines, metabolites and gut microbiome. Participants will complete patient reported outcomes (PROs) weekly. The investigators will collect fasting labs and research blood with each cycle of chemotherapy (4 instances). The investigators will also collect research bloods at baseline. The investigators will collect stool samples at baseline, and after fasting interventions for Cycle 1 and 3.

Through the proposed investigations the investigators will test the feasibility of a promising strategy to augment delivery of chemotherapy in a population at risk for toxicity for cancer therapy, and explore the mechanisms by which it may function. The long-term goals are to: enhance patient experience during chemotherapy, improve survival outcomes, and reduce disparities in survival between those who received recommended dose of chemotherapy versus those who require a dose reduction due to side effects. The study can potentially move the field forward by (a) identifying key cytokine, microbiome and metabolome changes associated with short-term fasting in ESBC and (b) improving survival outcomes in patients with ESBC.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with histologically-confirmed stage I-III invasive carcinoma of the breast
* Planning for standard neoadjuvant or adjuvant chemotherapy ddAC or TC for 4 cycles (concurrent anti-HER2 therapy is permitted)
* Provider physical exam within 4 weeks of consent
* Eastern Cooperative Oncology Group (ECOG) 0-1 (as per recent provider note or direct confirmation with provider)
* BMI ≥ 19.5 kg/m2 (as per most recent visit documented in medical record)
* Willingness to change diet, and provide fecal sample 3 times during study

Exclusion Criteria:

* BMI <19.5 kg/m2
* Diabetes
* History of eating disorder
* Serious/uncontrolled medical condition (e.g. end stage renal disease on dialysis, cirrhosis, uncontrolled hypertension, seizure disorder, history of bariatric surgery)
* Pregnant or nursing
* Use of medications that must be taken with food: allopurinol, aspirin, amiodarone, baclofen, bromocriptine, carvedilol, carbamezpine, cimetidine, diclofenac, doxycycline, fenofibrate, fludrocortisone, glyburide, hydrocortisone, iron supplements, ketorolac, lithium, methylprednisolone, naproxen, niacin, potassium salts, prednisone, procainamide, sevelamer, sulfasalazine, trazodone, valproic acid

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women with early stage breast cancer (HER2-negative) planning to receive chemotherapy
Enrollment: 30 (Estimated)
Dates: Start 2024-08-08 (Actual); Primary Completion 2028-08 (Estimated); Study Completion 2029-05 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with self-reported adherence to the fasting regimen | 6 -8 months
  Determine the feasibility of water-only fasting during chemotherapy in patients with invasive ESBC receiving cytotoxic chemotherapy.

SECONDARY OUTCOMES:
Rate of high-grade adverse effects | 6-8 months
  Evaluate the rate of any high-grade adverse effects (severe/very severe) during chemotherapy
Rate of Hematologic Toxicities | 6-8 months
  Evaluate the rate of high-grade hematologic toxicities during chemotherapy
Number of Dose Reductions or Dose Delays | 6-8 months
  Evaluate the total number of dose reductions or delays
Percent Change in Quality of Life Questionnaire The European Organisation for Research and Treatment Cancer C30 score | 6 months, 12 months
  Participants will complete the Quality of Life Questionnaire C30 The Quality of Life Questionnaire-C30, which includes 30 items. The 30 items assess physical, role, emotional, cognitive and social functioning, global health status or Quality Of Life scales, fatigue, pain, nausea and vomiting, dyspnea, insomnia, appetite loss, constipation, diarrhea and financial difficulties. The Quality of Life Questionnaire-C30 is scored on the basis of classical test theory (CTT), and uses the total item score as the scale score. All of the scales and single-item measures range in score from 0 to 100. Higher score for the functioning scales and global health status denote a better level of functioning (i.e. a better state of the patient), while higher scores on the symptom and single-item scales indicate a higher level of symptoms (i.e. a worse state of the patient). The percent change in Patient Reported Outcome scores from baseline is accessed at 6 and 12 months.
Percent change in Functional Assessment of Chronic Illness Therapy-Fatigue Scale | 6 months, 12 months
  Participants will complete the Functional Assessment of Chronic Illness Therapy-Fatigue Scale (FACIT-Fatigue) which includes 13 items. The 13 items assess self-reported fatigue and its impact upon daily activities and function. Response scale is 5 point Likert-type scale with manual scoring template, some items are reverse scored. Scale range is 0 to 52 with O being most fatigue and 52 indicating no fatigue. The percent change in fatigue scores from baseline is accessed at 6 and 12 months.
Changes in Key Inflammatory Cytokines/Chemokines | Baseline, 6-8 months
  Compare changes in key inflammatory cytokines/chemokines (IL4, IL6, IL22, IL17, CXCL5, and CXCL11), adipokines (Leptin, Adiponectin, Lipocalin, retinol-binding protein 4 (RBP4), Resistin, Ghrelin, and Omentin) from baseline to after each fast
Compare Changes in Tumor Cells | Baseline, 6-8 months
  Compare changes in tumor cells (AMPK, TSC1/2, STK11, mTOR) and intratumoral b-hydroxybutyrate from baseline to after each fast (if receiving neoadjuvant chemotherapy)
Compare Modulation of Gut Microbiome | Baseline, 6-8 months
  Examine the modulation of gut microbiome in response to fasting (for cycles 1 and 3) and compare it to baseline composition.
Compare the Composition of Gut Microbiome | Baseline, 6-8 months
  Compare the composition of the gut microbiome from baseline to after fasting (for Cycles 1 and 3) in individuals whose labs are consistent with fasting versus individuals whose labs are inconsistent with fasting (elevated b-hydroxybutyrate, low insulin, glucose and insulin like growth factor 1 (IGF-1))

OTHER OUTCOMES:
Absolute Percentage Change in Ki-67 | Pre neoadjuvant chemotherapy, post neoadjuvant chemotherapy up to 2 years
  Compare the absolute percentage change in Ki-67 and pathologic complete response prior to and following neoadjuvant chemotherapy
Prevalence of AA Genotype | 1-2 years
  Assess prevalence of AA genotype of MnSOD in patient with early stage breast cancer and if a greater proportion of women with the AA genotype have fewer side effects and improvement in biomarkers after fasting compared to the women who do not.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Sheng, MD, Principal Investigator — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (1):
- Sibley Memorial Hospital, Washington D.C., District of Columbia, United States